CLINICAL TRIAL: NCT01842503
Title: A Phase 1b/2a, Cross-over, Randomised, Double-blind, Placebo Controlled Study to Investigate the Safety and Pharmacodynamic Effects of GET 73 in Alcohol Dependent Subjects
Brief Title: Safety and Pharmacodynamic Study of GET 73 in Alcohol Dependent
Acronym: SPAD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Laboratorio Farmaceutico Ct S.r.l. (Industry)
Collaborators: Voisin Consulting, Inc. (Industry); Latis S.r.l. (Industry); Quotient Bioresearch (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 73CT-2-03; 2012-005515-13 (EudraCT Number)
Record Dates: First submitted 2012-12-20; First posted 2013-04-29 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Alcohol Dependence
Keywords: alcohol dependence; cue reactivity; alcohol self administration
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GET 73 (Active Comparator): 300 mg (3 capsules) tid for 3 days
  Interventions: Drug: GET 73
- inactive ingredients capsule (Placebo Comparator): 3 capsules tid for 3 days
  Interventions: Drug: inactive ingredients capsule

INTERVENTIONS:
Drug: GET 73 — 300 mg tid on 3 days cycle
  Arms: GET 73
Drug: inactive ingredients capsule — 3 capsules tid on 3 days cycle
  Arms: inactive ingredients capsule

SUMMARY:
Examination of the effect of GET 73 on alcohol pharmacokinetics and pharmacodynamics (intoxication and sedation)and safety profile in alcohol-dependent individuals.To evaluate whether GET 73, as compared to placebo, results in diminished cue-reactivity responses to alcohol cues in terms of urge to drink during the cue reactivity session and results in lower quantity of alcohol consumed during an alcohol self-administration session.

ELIGIBILITY:
Inclusion Criteria:

* male or female subjects, between 21 and 65 years old (inclusive);
* participants must meet criteria for current Diagnostic and Statistical Manual (DSM-IV)diagnosis of alcohol dependence,supported by the structured clinical interview for DSM-IV Axis I Disorders Patient Edition;
* participants must meet criteria for heavy drinking, defined as averaging

  * 4 drinks/day for women and ≥5 drinks/day for men during a 30-day period within the 90 days prior to screening evaluation;
* participants must be in good health as confirmed by medical history, physical examination, ECG, lab tests;
* females must be postmenopausal for at least one year or surgically sterile. Otherwise, females will be excluded (even if they are using any kind of birth control). Proof (medical records, certification from an medical doctor) of surgical sterility will be required. Certification of postmenopausal for at least 1 year and postmenopausal levels of FSH will also be required to be into the study;
* participants must be willing to take oral medication and adhere to the study procedures;
* participants must give their consent to enter the study by signing the informed consent form.

Exclusion Criteria:

* individuals seeking treatment for alcohol dependence;
* positive urine drug screen at baseline for positive drug screen for the following: opioids, benzodiazepines, cocaine, methamphetamine or any other stimulants. A urine drug screen may be repeated once and must test negative before randomization;
* individuals diagnosed with a current substance dependence, other than alcohol or nicotine;
* meet DSM-IV Axis I criteria for a lifetime diagnosis of schizophrenia, bipolar disorder, or other psychoses;
* Subjects taking any psychoactive medication that in the opinion of the subjects primary care physician, cannot be discontinued at least 14 days prior to being randomized;
* an active illness within the past 6 months of Visit 1 that meet the DSM-IV criteria for a diagnosis of Major Depressive Disorder or Anxiety Disorder;
* subjects with a history of suicide attempts and/or at risk for suicide will be excluded, based on the Structured Clinical Interview Disorders assessment and on the Investigators' evaluation;
* clinically significant medical abnormalities (i.e., unstable hypertension, clinically significant abnormal ECG, bilirubin > 150% of the upper normal limit, alanine aminotransferase or aspartate aminotransferase elevations >300% the upper normal limit, estimated creatinine clearance ≤ 60 dl/min);
* current use of any medications prescribed to reduce alcohol use e.g. naltrexone, acamprosate, disulfiram or topiramate;
* concomitant use of cytochromeP450 2C19 substrates; assumption of cytochromeP450 2C19 and cytochromeP450 3A4 inhibitors or inducers in the 14 days before dosing;
* individuals with a reasonable expectation of being institutionalized during the course of the trial;
* participants who have significant alcohol withdrawal symptoms, defined as a Clinical Institute Withdrawal Assessment >10;
* history of seizures (e.g. epilepsy), including alcohol-related seizures;
* history of delirium tremens;
* subjects who have participated in any behavioral and/or pharmacological study within the past 30 days;
* history of delirium tremens.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
changes in area under the plasma concentration of alcohol versus time curve (AUC), after administration of GET 73 or placebo | blood samples are drawn on day 2 and day 12 at baseline and then, following the start of alcohol consumption, for the next 8 hours or until the blood alcohol level is zero on 2 successive determinations
  On Day 2 and Day 12 subjects have an indwelling catheter placed in a forearm vein for blood draws. After the 5th dose of GET 73 or placebo is administered on Day 2 and Day 12, participants receive a dose of alcohol 30 minutes later, which is calculated to produce a peak of 0.08 g/L, based on body water content.
  AUC will be evaluated as mean value of overall subjects evaluated
Changes in pleasurable and negative effects of alcohol intoxication and sedation, measured by the Biphasic Alcohol Effects Scales (BAES),during the Alcohol Self-Administration (ASA) session, when taking GET 73 compared to placebo. | The BAES will be administered, at Day 2 and Day 12, eight times after the priming drink is presented during the ASA.
Changes in reaction time, measured by Conners's Continuous Performance Task (CPT),when taking GET 73 compared to placebo | CPT will be assessed at Day 2 and Day 12
Changes in cognitive performance, measured by Digit Symbol Substitution Test (DSST), when taking GET 73 compared to placebo | DSST will be assessed at Day 2 and Day 12
Frequency of adverse events (AEs) occured after placebo or GET 73 administration | up to 20-27 days
  All AEs occurring during the study will be recorded. Subjects are discharged from the hospital at Day 13, after the two inpatient treatment phases (Day 1-Day 3 and Day 11-Day 13). A follow-up visit, approximately from 7 to 14 days after the second CR/ASA experiment, will be performed. The AEs will be grouped by Medical Dictionary for Regulatory Affairs preferred terms into frequency tables according to system organ class (SOC).
  Frequencies of AEs occurred after placebo or GET 73 administration will be compared using chi-square or Fischer's exact test.
Changes in cue reactivity (CR) responses to alcohol cues, in terms of urge to drink, as measured by the Alcohol Urge Questionnaire (AUQ), when taking GET 73 compared to placebo. | At Day 3 and Day 13 during the two treatment phases
  To evaluate whether GET 73, as compared to placebo, results in reductions in craving (as measured by the AUQ), the AUQ will be administered eight times after the priming drink is presented during the ASA.
Changes in CR responses to alcohol cues, in terms of psychophysiological responses,heart rate,mean arterial pressure and salivation changes during the CR session. | At Day 3 and Day 13 during the two treatment phases
  There are three experimental time periods of 3-minutes each during each CR session. Cotton swabs will be weighed at the end of each 3-minute block and the mean values for weight of salivation will be calculated. An average heart rate and an average mean arterial pressure will be calculated for each of these three time periods.
Changes in attention to the sight and smell of cues, as measured by Alcohol Attention Scale (AAS), during the CR. | This endpoint will be measured twice in each CR session (Day 3 and Day 13) through the AAS.
Effects of GET 73 on the amount of alcohol consumed during the ASA. The maximum quantity of alcohol will be taken, to have a measure directly comparable to AUQ results | At Day 3 and Day 13 during the two treatment phases
Changes in peak plasma concentration (Cmax) of alcohol after administration of GET 73 or placebo | blood samples are drawn on Day 2 and Day 12 at baseline and then, following the start of alcohol consumption, for the next 8 hours or until the blood alcohol level is zero on 2 successive determinations
  Cmax will be calculated at the peak level as mean value of overall subjects evaluated
Changes in time to peak plasma level (Tmax) of alcohol after administration of GET 73 or placebo | blood samples are drawn on Day 2 and Day 12 at baseline and then, following the start of alcohol consumption, for the next 8 hours or until the blood alcohol level is zero on 2 successive determinations
  Tmax will be evaluated as the time after administration corresponding to the time of peak plasma level and as mean value of overall subjects evaluated
Changes in half-life of alcohol after administration of GET 73 or placebo | blood samples are drawn on Day 2 and Day 12 at baseline and then, following the start of alcohol consumption, for the next 8 hours or until the blood alcohol level is zero on 2 successive determinations
  Half-life will be calculated as mean value of overall subjects evaluated
Characteristics of adverse events (AEs) occured after placebo or GET 73 administration | up to 20-27 days
  All AEs occurring during the study will be recorded. Subjects are discharged from the hospital at Day 13, after the two inpatient treatment phases (Day 1-Day 3 and Day 11-Day 13). A follow-up visit, approximately from 7 to 14 days after the second CR/ASA experiment, will be performed. The AEs will be grouped by Medical Dictionary for Regulatory Affairs preferred terms according to system organ class (SOC). When an AE occurs more than once for a subject, the maximal severity and strongest relationship to the medication will be counted.
  Characteristics of AEs occurred after placebo or GET 73 administration will be compared using chi-square or Fischer's exact test.

CONTACTS AND LOCATIONS:
Overall Officials: Robert M. Swift, M.D., R.Ph., Principal Investigator — Roger Williams Medical Center
Locations (1):
- Roger Williams Medical Center, Providence, Rhode Island, United States